CLINICAL TRIAL: NCT02845089
Title: Treatment Patterns, Outcomes and Resource Use Study for Advanced Stage Non-Small Cell Lung Cancer (Squamous and Non-squamous) in the Kingdom of Saudi Arabia and United Arab Emirates
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-454
Record Dates: First submitted 2016-07-08; First posted 2016-07-27 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced/Metastatic NSCLC patients from UAE and KSA: A random sample of patients diagnosed with advanced/metastatic non-small cell lung cancer (NSCLC) from select oncology centers in Kingdom of Saudi Arabia (KSA) and United Arab Emirates (UAE)

SUMMARY:
A retrospective observational longitudinal medical chart review study of randomly sampled patients diagnosed with advanced/metastatic NSCLC. The minimum observational period for each patient will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older at the time of advanced/metastatic NSCLC diagnosis, and currently alive or deceased
* Histologically confirmed diagnosis of advanced/metastatic NSCLC (squamous, non-squamous or NOS) stages IIIB/IV. First diagnosis of advanced/metastatic NSCLC between 01-Jan-2010 and 31-Mar-2014 (currently alive or deceased) with a minimum 12 months of potential observation period available in medical records
* Medical history and treatment data must be available (or obtainable by SI) for chart abstraction from the date of advanced/metastatic diagnosis through most recent patient follow-up/contact. This also includes documentation of treatment by other physicians and inpatient hospital treatments within KSA or the Health Authority of Abu Dhabi (HAAD) system
* Patients must have at least all data on age, gender, date of advanced NSCLC diagnosis, Line of Treatment (LOT) information (agent types and dosage), and date of last follow-up

Exclusion Criteria:

* Patient had enrolled in a cancer treatment-related clinical study at any time after the diagnosis of advanced/metastatic NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A random sample of patients diagnosed with advanced/metastatic NSCLC from select oncology centers in UAE and KSA
Sampling Method: Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Patient Demographics at diagnosis with advanced/metastatic NSCLC | at baseline
Systemic treatments prescribed for NSCLC patients from treatment initiation through discontinuation | approximately 12 months
Duration of systemic treatments | approximately 12 months
Distribution of reasons for discontinuing treatment | approximately 12 months

SECONDARY OUTCOMES:
healthcare resource utilization in patients with advanced/metastatic NSCLC | approximately 12 months
  NSCLC-related health care resources associated with the provision of systemic treatments and managing side effects of treatments: hospital admissions including emergency room visits
Progression-Free Survival (PFS) | approximately 12 months
Overall Survival (OS) | approximately 12 months
Adverse Events (AEs) | approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx